CLINICAL TRIAL: NCT06918236
Title: Association of Assisted Reproductive Technologies Parameters With the Perinatal Outcome in Singleton and Multiple Pregnancies: A Multicenter Prospective Cohort Study
Brief Title: Association of Assisted Reproductive Technologies Parameters With the Perinatal Outcome
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Hospital Universitario de Torrejón,Madrid (Other); Universidad Francisco de Vitoria (Other); University Hospital, Pleven, Bulgaria (Unknown); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Universitario de Canarias (Other)
Responsible Party: Principal Investigator, Themistoklis Dagklis, Associate Professor of Obstetrics and Gynecology, Aristotle University Of Thessaloniki
Other Study IDs: 320/2024
Record Dates: First submitted 2025-03-29; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Fetal Growth Restriction (FGR); Preeclampsia; Stillbirth; Placenta Previa; Vasa Previa; Small for Gestational Age (SGA)
Keywords: fetal growth restriction; Preeclampsia; stillbirth; placenta previa; vasa previa; Assisted reproductive techniques; ART; Small for Gestational Age (SGA); IVF; ICSI
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia; Stillbirth; Placenta Previa; Vasa Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ART group - Study group: The study group will include pregnant individuals aged 18 years or older with singleton or multiple pregnancies conceived through assisted reproductive technologies. Participants will be recruited during routine first-trimester ultrasound examinations between 11 weeks plus 0 days and 13 weeks plus 6 days of gestation at participating fetal medicine units. Pregnancies with major fetal anomalies or known genetic conditions will be excluded from the primary analysis.
- Natural conception group- Control group: The control group will include pregnant individuals aged 18 years or older with singleton or multiple pregnancies conceived spontaneously, without the use of assisted reproductive technologies. Participants will be recruited during routine first-trimester ultrasound examinations between 11 weeks plus 0 days and 13 weeks plus 6 days of gestation at participating fetal medicine units. Pregnancies with major fetal anomalies or known genetic conditions will be excluded from the primary analysis.

SUMMARY:
The goal of this prospective cohort study is to examine how different parameters of assisted reproductive technologies (ART) are associated with the perinatal outcome in individuals with singleton or multiple gestations. The main questions it aims to answer are:

Are ART pregnancies associated with a higher risk of:

* Small for gestational age neonates?
* Fetal growth restriction, either early- or late-onset?
* Development of preeclampsia?
* Stillbirth (intrauterine fetal death after 22 weeks not due to known anomalies)?
* Are certain ART parameters-such as the type of fertilization (e.g., IVF vs. ICSI), embryo stage at transfer, use of fresh vs. frozen embryos, or ovarian stimulation protocols-more strongly associated with adverse outcomes?

Are ART pregnancies associated with placental and umbilical cord abnormalities, including:

* Placenta previa?
* Vasa previa?
* Single umbilical artery?
* Velamentous or marginal cord insertion?

Researchers will compare outcomes between pregnancies conceived through ART and those conceived spontaneously.

Participants will:

* Be individuals aged 18 or older undergoing routine first-trimester ultrasound between 11 and 14 weeks of gestation
* Provide detailed medical, obstetric, and ART-related information
* Undergo routine prenatal assessments, including ultrasound evaluations of fetal growth, Doppler studies, and placental characteristics
* Have perinatal outcomes such as gestational age at birth, mode of delivery, birthweight, and complications systematically recorded

Statistical models will be used to adjust for confounding factors such as maternal age, BMI, parity, and smoking.

The aim is to better understand how ART and specific ART parameters may influence maternal and neonatal health and to improve counseling and clinical care for people using fertility treatments.

DETAILED DESCRIPTION:
Rationale:

In this multicenter prospective cohort study, our primary aim is to determine the association of various assisted reproductive technologies (ART) parameters with the perinatal outcome after adjusting for key confounders such as maternal age, BMI, parity and smoking. Our primary outcomes will be small for gestational age neonates, fetal growth restriction, preeclampsia and stillbirth. Additionally, the investigators will examine the association between ART and a range of placental/umbilical abnormalities-such as placenta previa, vasa previa, single umbilical artery, and abnormal cord insertions-and explore how these structural aberrations may act as a mediator. Together, this comprehensive approach is intended to clarify the mechanisms linking ART to adverse obstetric outcomes and ultimately inform improved clinical care and counseling for couples considering ART.

Objectives:

Primary Objective:

To evaluate the association between ART parameters and a series of adverse perinatal outcomes both in singleton and in multiple pregnancies, analyzed as distinct populations. ART pregnancies will be examined both as a collective cohort and within subgroups stratified by specific ART techniques and treatment protocols.

Our primary outcomes under investigation:

* Small for gestational age neonates defined as <10th percentile.
* Fetal growth restriction, either early-onset (<32 weeks) or late-onset (>32 weeks), characterized by an estimated fetal weight below the 3rd percentile or below the 10th percentile based on the Fetal Medicine Foundation (FMF) fetal growth charts accompanied by abnormal Doppler findings; or birthweight below the 5th centile based on the FMF neonatal growth charts
* Development of preeclampsia
* Stillbirth (intrauterine demise after 22 weeks gestation not attributable to other causes (i.e. congenital infections, structural defects, genetic anomalies)

Secondary Objectives:

To investigate the relationship between ART and various placental as well as umbilical cord abnormalities (e.g., placenta previa, vasa previa, single umbilical artery, velamentous and marginal cord insertions).

All analyses will be adjusted for maternal age, BMI, parity, smoking and other significant confounders depending on the investigated outcome.

Methods and analysis:

Design, participants and timeframe of enrollment and visits:

The study will be a prospective observational cohort that will include all consecutive women above 18 years old who attend for routine ultrasound examination at 11+0 to 13+6 weeks of gestation at one of participating fetal medicine units. The eligibility criteria will be: singleton or multiple pregnancies, with a live fetus at 11+0 to 13+6 weeks, without known genetic anomalies or major fetal defects (such as acrania, holoprosencephaly, megacystis, exomphalos, congenital heart defects) diagnosed before or after birth. All sonographers will be certified for the first-trimester scan by the FMF. Approval will be secured from the ethical committee at each participating center. In every case, written informed patient consent will be obtained.

During the initial consultation, maternal height, weight and sociodemographic details such as maternal age, parity, smoking and procedure details in cases of ART conception will be recorded. Detailed demographic information, individual, obstetric, and family history, as well as any complications during the current pregnancy, will be systematically recorded. At each prenatal visit, the investigators will document obstetric ultrasound findings-including fetal growth percentiles, amniotic fluid index, and Doppler measurements-following all protocols recommended by the FMF relevant to the case.

Collection of ART Methodology Data:

Taking into account our objective, to conduct a detailed analysis of each ART method and parameter in relation to the perinatal outcome, including subgroup analyses based on specific techniques and protocols, the investigators will collect detailed information on ART methods and protocols using a standardized data collection form, which will include the following variables:

* Subfertility details: Type of subfertility (primary or secondary) and duration of subfertility. The investigators will document whether the subfertility is due to female factors, male factors, or both. Occurrence of ovarian hyperstimulation syndrome, categorized as mild, moderate or severe will also be recorded, particularly in fresh transfer cycles.
* Gamete origin: Source of sperm and oocytes, specifying whether they are from the same individual (autologous) or from a donor. The investigators will also note if the oocytes are fresh or frozen and the donor age.
* Culture conditions and media: Details about the embryonic culture environment, including whether an oxygen gradient was used or other specific culture media conditions, will be collected to assess their potential impact on embryo development.
* Type of fertilization: The method of fertilization employed, such as conventional IVF or intracytoplasmic sperm injection, will be documented.
* Embryo stage at transfer: The developmental stage of embryos at the time of transfer will be recorded, distinguishing between cleavage-stage embryos (day 2-3) and blastocyst-stage embryos (day 5).
* Type of embryo transferred: The investigators will specify whether fresh or frozen embryos were transferred during the procedure.
* Preimplantation Genetic Testing (PGT): Information on whether preimplantation genetic testing was performed will be collected, including the timing of the testing (day 3 or day 5) and the type of testing, together with any other prenatal or postnatal genetic testing.
* Embryo details: The number of embryos available and the number transferred will be noted. The classification and quality of embryos based on morphological and genetic assessments will be recorded. If mosaic embryos were transferred, the investigators will document the levels of mosaicism and any instances of confined placental mosaicism together with any other prenatal or postnatal genetic testing.
* Stimulation Protocol: Details of the ovarian stimulation protocol used will be collected, including whether a gonadotropin-releasing hormone (GnRH) antagonist protocol, GnRH agonist long protocol, GnRH agonist short protocol, or GnRH agonist ultra-short protocol was employed.

Monitoring and Follow-up:

Throughout the pregnancy, any complications such as growth disorders, preeclampsia, stillbirth, gestational diabetes, hypertensive disorders, placental abruption, preterm premature rupture of membranes and spontaneous preterm labor will be closely monitored and recorded. Detailed ultrasonographic assessments of placental and umbilical cord abnormalities (e.g., cord insertion site, number of vessels, placental location) will be performed and recorded, together with details on direct examination at birth and any prenatal or postnatal genetic testing, if available. Even though cases with known genetic anomalies or major fetal defects will be excluded from our primary and secondary analyses, the investigators will systematically record fetal structural anomalies, aneuploidies, and congenital defects based on prenatal ultrasonographic assessments and confirmed postnatally whenever applicable, including findings from genetic testing and direct neonatal examination.

Obstetric ultrasound findings, including fetal growth percentiles, amniotic fluid index, and Doppler indices, will be documented at each visit. Following delivery, perinatal outcomes such as gestational age at birth, onset of labor (spontaneous rupture of membranes, contractions, induction, or elective cesarean section), mode of delivery (vaginal or cesarean), birth weight and birth weight percentile according to FMF neonatal percentiles, Apgar scores, and postpartum complications (e.g., postpartum hemorrhage) will be recorded.

Data collection:

An electronic case record form (CRF) has been specifically designed for this study and incorporated into the clinical software used at the participating centers (ViewPoint® software, GE Healthcare; Munich, Germany or Astraia© software, NEXUS / ASTRAIA GmbH, Ismaning, Germany). Data will be entered prospectively during the study. Access to data included in the CRF will be restricted to the investigators involved in each participating site.

Recruitment and power-sample size estimation:

For the power analysis, the investigators chose the rarer outcome among our primary outcomes, stillbirth. A relevant prospective cohort reported that the prevalence of stillbirth is 3.7‰ among singleton pregnancies that were conceived naturally, while the risk of stillbirth among IVF-ART pregnancies was 16.2‰. To detect such an increase with a statistical power of 0.80 and a significance level of 0.05, at least 989 ART pregnancies will be needed. After adjusting for a 1:10 ratio of ART pregnancies to spontaneous conceptions, based on data from our study population in previous research, and increasing the sample size by 10% to account for potential losses during follow-up, the investigators determined a required sample size of 1,099 study cases and 10,985 control pregnancies, for a total of 12,084 pregnancies.

Data management and statistical analyses:

Singleton and multiple pregnancies will be investigated as separate populations. The pregnancies resulting from ART will serve as the study population, while pregnancies from spontaneous conception will form the control group. For every investigated outcome multivariate logistic regression analyses will be conducted, incorporating ART use as an independent variable along with available potential confounding factors. For each analysis, essential confounders will include maternal age, BMI, parity and smoking, while other confounders will be considered based on the individual dependent variable being examined and the decision to include them will be based on clinical relevancy.

In addition to multivariate logistic regression, propensity score matching will be employed as a sensitivity analysis for the statistically significant outcomes to further account for confounders. Using the R programming language, the investigators will create propensity scores based on the same confounders used in the logistic regression analyses for each specific outcome. Participants in the ART group will be matched to participants in the spontaneous conception group based on their propensity scores and the balance will be assessed using the standardized mean differences. This matching process aims to balance the distribution of confounders between the two groups, thereby reducing selection bias and providing an alternative estimation of the effect of ART on the outcomes of interest. After matching, statistical tests appropriate for paired data will be employed, depending on the investigated association, as suggested by relevant literature.

When feasible, subgroup analyses will be performed to investigate the effects of different ART methods and parameters on the investigated outcomes.

The investigators will examine missing data fields to identify the type of missing data mechanisms. Due to the type of outcomes studied, the investigators believe that the majority of missing data will be missing at random; thus, as a sensitivity analysis, multiple imputation technique will be used to impute the missing data. If there are informatively missing data due to clinically relevant events such as death or critical illness the investigators will examine statistical models to account for missing not at random.

Adjusted odds ratios and 95% confidence intervals will be calculated for all analyses. A statistical significance level of 0.05 will be applied. All analyses will be performed using the R programming language.

ELIGIBILITY:
Inclusion Criteria

* Singleton or multiple pregnancies
* Live fetus between 11 weeks plus 0 days and 13 weeks plus 6 days of gestation

Exclusion Criteria

* Known genetic anomalies diagnosed before or after birth
* Major fetal defects diagnosed before or after birth, such as acrania, holoprosencephaly, megacystis, exomphalos, congenital heart defects

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive women 18 years old or older who attend for routine ultrasound examination at 11 weeks plus 0 days to 13 weeks plus 6 days of gestation at one of participating fetal medicine units.
Sampling Method: Non-Probability Sample
Enrollment: 12084 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Small for gestational age neonates | At delivery/birth
  Small for gestational age neonates defined as birthweight lower than the 10th percentile
Development of preeclampsia | From the 20th gestational week and up to 8 weeks after the delivery/birth
  New onset of hypertension (systolic pressure ≥140 and/or diastolic pressure ≥90 mmHg) and proteinuria or the new onset of hypertension plus significant end-organ dysfunction with or without proteinuria, typically presenting after 20 weeks of gestation or postpartum.
Fetal growth restriction | From the 22nd gestational week and up to the delivery/birth
  Fetal growth restriction, either early-onset (<32 weeks) or late-onset (>32 weeks), characterized by an estimated fetal weight below the 3rd percentile or below the 10th percentile based on the Fetal Medicine Foundation fetal growth charts accompanied by abnormal Doppler findings; or birthweight below the 5th centile based on the FMF neonatal growth charts
Stillbirth | From the 24th gestational week and up to the delivery/birth
  Stillbirth (intrauterine demise after 22 weeks gestation not attributable to other causes (i.e. congenital infections, structural defects, genetic anomalies)

SECONDARY OUTCOMES:
Placenta previa | From the 20th gestational week up to the 24th gestational week.
  Placenta partially or completely covers the internal cervical os.
Vasa previa | From the 20th gestational week up to the 24th gestational week.
  Vasa previa occurs when fetal blood vessels that are unprotected by the umbilical cord or placenta run through the amniotic membranes and traverse the cervix.
Single umbilical artery | From the 20th gestational week up to the 24th gestational week.
  Umbilical cord with one instead of two umbilical arteries
Velamentous and marginal cord insertions | From the 20th gestational week up to the 24th gestational week.
  Abnormal cord insertions

CONTACTS AND LOCATIONS:
Locations (6):
- University Hospital of Pleven, Pleven, Bulgaria
- Aristotle University of Thessaloniki, Thessaloniki, Central Macedonia, Greece
- Spain (4):
  - Complejo Hospitalario Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Universidad Francisco de Vitoria, Madrid
  - Hospital Universitario de Torrejón, Madrid
  - Hospital Clínico Universitario "virgen de la Arrixaca", Murcia